CLINICAL TRIAL: NCT05365009
Title: Characteristics of Patients With Autoimmune Interstitial Lund Disease From Argentina
Brief Title: Registry of Autoimmune Interstitial Lung Disease
Acronym: EPIMAR
Status: Recruiting | Type: Observational
Sponsor: EPIMAR registry (Network)
Collaborators: Sociedad Argentina de Reumatologia (Other)
Responsible Party: Sponsor
Other Study IDs: 2022
Record Dates: First submitted 2022-03-09; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Interstitial Lung Disease Due to Systemic Disease
Keywords: connective tissue disease; interstitial lung disease; rheumatoid arthritis; systemic sclerosis; interstitial penumonia with autoimmune features
MeSH Terms: conditions — Connective Tissue Diseases; Lung Diseases, Interstitial; Arthritis, Rheumatoid; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EPIMAR group: EPIMAR (ARgentina's Autoimmune Mechanism Interstitial Pulmonary Disease) registry was created in 2016 by a group of multidisciplinary specialists with experience in the management of ILD.
  Interventions: Diagnostic Test: Multidisciplinary aproach

INTERVENTIONS:
Diagnostic Test: Multidisciplinary aproach — regular tests

SUMMARY:
Interstitial lung diseases (ILD) constitute a group of entities characterized by inflammation and/or fibrosis of the lung parenchyma.

In recent years, with the advent of new diagnostic tools and therapeutic options, multidisciplinary evaluation is essential, since it optimizes the interpretation of each case and the quality of care for these pathologies Consensus for the identification and management of ILD associated with SSc (ILD-SSc) is the only guideline published at present. In the others autoimmune ILD (Ai-ILD), screening, diagnosis, treatment and follow-up strategies are usually performed according to the criteria of the treating medical team. Guidelines regarding the follow-up and indication of immunosuppressive and antifibrotic treatment are lacking. Many questions on the horizon of the Ai-ILD should be answered as better quality evidence emerges from studies with a greater number of patients and better methodological design.

DETAILED DESCRIPTION:
Autoimmune ILD (Ai-ILD) include ILD associated with connective tissue disease (CTD), ILD associated with antineutrophil cytoplasmic antibodies (ANCA-ILD) and interstitial pneumonia with autoimmune findings (IPAF).

PRIMARY OBJECTIVE To describe the baseline sociodemographic, clinical, serological, functional, radiological and treatment characteristics of patients with Ai-ILD and in the 5-year follow-up.

GENERAL OBJECTIVES

1. To know the frequency of subclinical Ai-ILD and its evolution.
2. To identify risk factors associated with the progression of Ai-ILD.
3. To characterize the subgroup of patients with progressive fibrosing phenotype.
4. To describe patterns of treatments used with Ai-ILD.
5. To describe the most frequent adverse drug events.
6. To evaluate global mortality and the factors associated with annual and 5-year survival.

SPECIFIC OBJECTIVES To characterize patients with ILD associated with each of the most common autoimmune diseases, ANCA-ILD and IPAF.

To describe the prescription patterns according to the underlying autoimmune entity and the severity of the ILD presentation.

To study the lung function changes in patients treated with immunosuppressants and / or antifibrotics.

To report adverse events and long-term safety associated with the use of different prescribed drugs.

To describe the survival of the treatments used. To know the accessibility to prescribed therapies. To know the frequency of use of health resources. To describe the impact of the disease on quality of life and work activity.

STUDY DESIGN The EPIMAR II registry will have a prospective, observational and multicenter design.

The inclusion of new patients for the follow-up cohort (EPIMAR II) will begin in 2021. Patients evaluated and diagnosed in the last 5 years who are currently under follow-up will be included. They will be evaluated at a baseline visit and then annually. Patients in the EPIMAR I cohort who meet the inclusion criteria may be included in this new registry.

POPULATION Patients with a diagnosis of Ai-ILD according to the evaluation of a multidisciplinary team. Patients without respiratory symptoms may be included in the registry and will be classified as subclinical ILD.

INCLUSION CRITERIA

* Age ≥ 18 years old
* Diagnosis of ILD within the last 5 years according to the criteria of the multidisciplinary team composed of at least one pulmonologist and one rheumatologist, with or without respiratory symptoms.
* ILD defined by the presence of ground glass opacities and / or peribronchovascular or airspace consolidations and / or reticulations and / or traction bronchiectasis and / or honeycomb on high-resolution computed tomography (HRCT) within the last 12 months
* One of the following three criteria:

Established or early stage CTD. IPAF according to ATS / ERS 2015 classification criteria. ANCA positivity by immunofluorescence confirmed by ELISA, with or without systemic vasculitis.

* Spirometry performed within the last 6 months before entering the registry.
* The participant must sign the informed consent voluntarily.

EXCLUSION CRITERIA Not being able to perform the clinical follow-up or the complementary studies required in the protocol.

Not being able to be evaluated by a multidisciplinary team; at least a rheumatologist plus a pulmonologist.

ILD associated with another non-autoimmune etiology according to the criteria of the multidisciplinary team (eg, occupational diseases, toxic)

RECRUITMENT

1. All rheumatologists and pulmonologists, members of SAR and AAMR will be invited to participate in the registry through scientific events, institutional emails, social networks, conferences.
2. The data will be collected into an online platform.
3. A multidisciplinary evaluation should be performed, considering a multidisciplinary team as a group of physicians from different specialties. The minimum requirement is at least a rheumatologist plus a pulmonologist. Other specialties (radiologists, pathologist, an internist with training and experience in autoimmune diseases) may also be part of this team.
4. Each research center will be compromised to perform the scheduled visits with the multidisciplinary evaluation requirements. The investigators will be selected and accepted by the EPIMAR coordinators.
5. To guarantee the homogeneity and quality of the information, each variable in the registry will have standardized definitions
6. The researchers will invite all consecutively patients that meet the inclusion criteria to participate in the registry.
7. Once the informed consent has been signed, a face-to-face interview will be performed in which the baseline information will be obtained and an exhaustive review of the patient's medical history will be developed.
8. Each patient to enter the registry must have a HRCT performed within 12 months and spirometry within the 6 months prior to the baseline visit.
9. A radiologist with 10 years of experience in thorax diseases will review the pulmonary images and will interpret and score each HRCT. The process will be centralized and blind
10. The investigator will conduct annual follow-up visits for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosis of ILD within the last 5 years according to the criteria of the multidisciplinary team composed of at least one pulmonologist and one rheumatologist, with or without respiratory symptoms.
* ILD defined by the presence of ground glass opacities and / or peribronchovascular or airspace consolidations and / or reticulations and / or traction bronchiectasis and / or honeycomb on high-resolution computed tomography (HRCT) within the last 12 months 17 .
* One of the following three criteria (see annex 1):

Established or early stage CTD 18-30. IPAF according to ATS / ERS 2015 classification criteria 8 ANCA positivity by immunofluorescence confirmed by ELISA, with or without systemic vasculitis 31.

* Spirometry performed within the last 6 months before entering the registry.
* The participant must sign the informed consent voluntarily.

Exclusion Criteria:

* Not being able to perform the clinical follow-up or the complementary studies required in the protocol.
* Not being able to be evaluated by a multidisciplinary team; at least a rheumatologist plus a pulmonologist.
* ILD associated with another non-autoimmune etiology according to the criteria of the multidisciplinary team (eg, occupational diseases, toxic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of ILD-Ai according to the evaluation of a multidisciplinary team. Patients without respiratory symptoms may be included in the registry and will be classified as subclinical ILD.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
  Number of patients that Survival at end of the study
Pulmonary test functionals | baseline and annual visits
  Change in functional tests over time (measurement of FVC and DLCO)
Fibrosis in Computed tomography | baseline and annual visits
  Change in Computed tomography in relation to fibrotic involvement, measured by the same operator

SECONDARY OUTCOMES:
Safety of the treatments used | 5 years
  number and type of event adverse

CONTACTS AND LOCATIONS:
Overall Officials: Florencia Vivero, MD, Principal Investigator — Sociedad Argentina Reumatologia
Locations (1):
- Epimar Ii, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: web site — http://www.arthrosoft.com/